CLINICAL TRIAL: NCT04109885
Title: Intramuscular Paracervical Injection for Headache in the Emergency Department: A Randomized Controlled Trial
Brief Title: Paracervical Injection for Headache in the Emergency Department
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Christian Fromm, MD (Other)
Responsible Party: Sponsor-Investigator, Christian Fromm, MD, Director of Clinical Trials, Albert Einstein Healthcare Network
Organization: Albert Einstein Healthcare Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-173
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Headache Disorders, Primary; Pain Management; Emergency Department
MeSH Terms: conditions — Headache Disorders, Primary; Agnosia; Emergencies | interventions — Prochlorperazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracervical injection (Experimental): 1.5 mL of 0.5% bupivacaine will be will be injected bilaterally in the paraspinal musculature of the cervical spine.
  Interventions: Drug: Paracervical injection
- Standard treatment (Active Comparator): Intravenous administration of prochlorperazine and diphenhydramine.
  Interventions: Drug: prochlorperazine and diphenhydramine.(Standard Treatment)

INTERVENTIONS:
Drug: Paracervical injection — 1.5 mL of 0.5% bupivacaine will be will be injected bilaterally in the paraspinal musculature of the cervical spine.
  Arms: Paracervical injection
Drug: prochlorperazine and diphenhydramine.(Standard Treatment) — Intravenous administration of prochlorperazine and diphenhydramine.
  Arms: Standard treatment

SUMMARY:
Headache is one of the most common presenting complaints in the emergency department.1 By the time patients with benign headaches present for treatment in the ED, they often have exhausted non-invasive treatments, and physicians are left with few therapeutic options. The investigators therefore propose to study the use of paracervical injection as a novel approach to managing headache in the emergency department. This procedure has great potential, if efficacious, to provide a safe, rapidly effective, non-sedating treatment for headache that does not involve intravenous line placement and systemic medication administration. To date, there are no published trials that evaluate this technique in this setting. The investigators intend to compare the efficacy of paracervical injection to standard first-line therapy (intravenous prochlorperazine and diphenhydramine) for the treatment of benign headache of any etiology in the emergency department.

DETAILED DESCRIPTION:
Headache is one of the most common presenting complaints in the emergency department.1 By the time patients with benign headaches present for treatment in the ED, they often have exhausted non-invasive treatments, and physicians are left with few therapeutic options.

Amongst the array of medications used by physicians to manage benign headache, dopamine antagonists have demonstrated the best efficacy in trials. A number of studies have demonstrated the efficacy of dopamine antagonists in treating migraine, tension, cluster-type, and other benign headaches2,3 Dopamine antagonists have shown superiority over opioids4, non-steroidal anti-inflammatory drugs5, triptans6, and anti-epileptics7. Prochlorperazine is probably the most studied and most commonly clinically utilized in this regard in the ED setting.

Despite the preponderance of evidence supporting the use of dopamine antagonists as first-line therapeutic agents in the ED management of benign headache, more than half of the 1.2 million patients treated in U.S. emergency departments for acute migraine are treated with opioids despite the known risks and recommendations to the contrary.12 In addition, there is tremendous variation in the medications chosen by ED physicians for managing benign headache.13 Most of these regimens involve administration of systemic medications that have considerable side effect profiles. Moreover, many of these headache cocktails require prolonged durations of treatment with sedative side effects. This results in prolonged ED lengths of stay that occupy valuable bed space in increasingly busy and crowded emergency departments.

A less well-known approach to managing benign headache is bilateral, paracervical, intramuscular injection of a long-acting anesthetic. The mechanism of action is not entirely understood, however it is postulated to involve neuronal pathways in the trigeminocervical complex thought to play a central role in headache physiology. This is similar in concept to the mechanism proposed for the occipital nerve blocks performed by neurologists.

Paracervical injection was first described by Mellick et al.8 This method has the advantage of ease of administration, favorable safety profile, lack of need for intravenous access, lack of sedative side effects, and swiftness of therapeutic response. In Mellick's case series, he treated 417 patients who presented with all manner of benign headaches with a 65% rate of complete relief of pain and a 20% rate of partial relief. Many patients had rapid relief of headache within 5 minutes and the remainder in less than 30 minutes. This study was limited by possible selection bias, given it is unclear why the specific patients enrolled were chosen for this treatment. The study was also limited by its observational nature and lack of a control group.

In recent years this procedure has gained popularity amongst emergency physicians, and it has been widely discussed in emergency medicine blogs and podcasts. Numerous online videos demonstrate the ease with which the procedure is performed by physicians and tolerated by patients. Many physicians have called for clinical trials to assess its efficacy.

The investigators therefore propose to study the use of paracervical injection as a novel approach to managing headache in the emergency department. This procedure has great potential, if efficacious, to provide a safe, rapidly effective, non-sedating treatment for headache that does not involve intravenous line placement and systemic medication administration. To date, there are no published trials that evaluate this technique in this setting. The investigators intend to compare the efficacy of paracervical injection to standard first-line therapy (intravenous prochlorperazine and diphenhydramine) for the treatment of benign headache of any etiology in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 64 years
* Suspected diagnosis of benign or primary headache

Exclusion Criteria:

* Treating attending physician is suspicious of a serious secondary cause of headache
* History of brain disease, concussion, stroke, intracranial mass or tumor, hemorrhage, increased intracranial pressure, head trauma in last 2 weeks, status post intracranial surgery
* History of neck disease, cervical spine or disc abnormality, history of vertebral or carotid artery dissection, torticollis, status post cervical spine surgery or hardware in place
* Hypersensitivity or allergy to bupivacaine (amide anesthetics) or prochlorperazine (dopamine receptor antagonists)
* Overlying signs of infection at site of injection (erythema, purulence, open skin)
* History of extrapyramidal symptoms, dystonia, parkinsonism, tardive dyskinesia or neuroleptic malignant syndrome
* Pregnancy
* History of schizophrenia or bipolar disorder
* Narcotic seeking patients as determined by the treating attending physician with optional assistance from medical record and online database review
* Weight more than 150 kg or less than 40 kg
* Received pain medication in the ED or less than 6 hours prior to enrollment
* Temperature greater than 38 degrees Celcius
* Previous enrollment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of symptom improvement | 30 minutes
  Patient asked if symptoms are improved enough for patient to be discharged to home.

SECONDARY OUTCOMES:
Reduction in pain scale | 30 minutes
  Pain scale measurement (1-10)
Re-presentation for medical care | 72 hours
  Patient asked if re-presented for medical care in the previous 72 hours (yes/no)
Headache recurrence | 72 hours
  Patient asked if headache recurred (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fromm, MD, Principal Investigator — Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No